CLINICAL TRIAL: NCT06374524
Title: Role of Greater Occipital Nerve Block in Headache From Spontaneous Intracranial Hypotension: a Prospective Observational Study
Brief Title: Greater Occipital Nerve Block for Spontaneous Intracranial Hypotension
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Anuj Bhatia, Professor, University Health Network, Toronto
Other Study IDs: 24-5568
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Spontaneous Intracranial Hypotension
MeSH Terms: conditions — Intracranial Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: greater occipital nerve block — Patients will receive an ultrasound-guided bilateral GONB (distal approach) of 5 mLs of injectate of bupivacaine 0.25% (5 mLs) + depomedrol 40 mg in 1 mL (3 mLs to each side).

SUMMARY:
Spontaneous Intracranial Hypotension (SIH) is a debilitating neurological disorder caused by a cerebrospinal fluid leak (CSF), with an estimated incidence of 5 per 100,000 persons per year, of which mostly women between the ages of 35 years and 55 years. The typical presentation is moderate-to-severe orthostatic headache and several other possible neurological symptoms, that significantly impact patients' quality of life.

Treatment of SIH usually starts with conservative measures, consisting of strict supine bed rest, hydration, caffeine, and simple analgesics. The vast majority of patients will require invasive treatments for their CSF leak, such as epidural blood patches, fibrin glue patches, endovascular coiling, and/or surgical repair. These specialized treatments are only offered in tertiary care centers and require specialized personnel and resources, which implicates a certain waiting time for the patients before permanent treatment is offered. In the meantime, due to the lack of an effective and accessible alternative, patients continue to suffer.

The greater occipital nerve block (GONB) has been reported as a simple, safe, and effective treatment to provide short-to-intermediate term relief of migraine, cervicogenic headache, cluster headache, occipital neuralgia, and more recently, post-dural puncture headaches (PDPH). As the pathophysiology of intracranial hypotension caused by SIH or PDPH is very similar, it is stipulated that the effect of GONB will be similar for SIH patients. However, to date, no studies exploring the efficacy of GONB for SIH have been performed.

The investigators propose to do a prospective observational study to explore the outcome of GONB for SIH. GONB can serve as a bridge therapy to control the debilitating headache of SIH while patients are awaiting permanent SIH treatment. Moreover, GONB can be performed by physicians of different specialties including neurology, which makes it an accessible treatment for all patients. Lastly, by offering better symptom control, this intervention could potentially restore patients' ability to work and reduce healthcare costs.

DETAILED DESCRIPTION:
This a prospective observational study on 34 patients with SIH, recruited from the Toronto Western Hospital Intracranial Hypotension Clinic. Patients will receive an ultrasound-guided bilateral GONB of 5 mls of injectate of mix of local anesthetic with steroid. There is no comparator. Primary outcome is the change in intensity of headache at 30 minutes post-intervention. Secondary outcomes are change in intensity up to day 14 post-intervention, onset of headache, sitting endurance, change in SIH-associated central nervous system (CNS) symptoms, emotional functioning, patient satisfaction, analgesic consumption and side-effect, up to 14 days post-intervention

ELIGIBILITY:
Inclusion criteria

1. Adults of > 18 years of age
2. Diagnosis of SIH, according to the International Classification of Headache Disorder (ICHD-3) classification (2)
3. Characteristics of pain:

   1. Baseline pain intensity NRS > 4/10 (in upright position)

Exclusion criteria

1. Contraindications to GONB: ongoing infection (systemic or located at the site of injection), intake of anticoagulants (not aspirin), allergy to injectate, contra-indication to injectate of steroids
2. Any significant cognitive or language barrier that impedes participation
3. Patients taking opioid medications with daily Oral Morphine Equivalent (OME) of 50 mg or higher
4. Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with documented SIH will be recruited from the Toronto Western Hospital Intracranial Hypotension Clinic and enrolled after consent is obtained.
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in headache intensity | 30 minutes post intervention
  The difference in the change in intensity of headache, as measured on an 11-point Numerical Rating Scale (NRS), measured 30 minutes after the intervention, after being positioned in an upright position for 10 minutes, compared to baseline.

SECONDARY OUTCOMES:
pain intensity | day 1,3,7,14
  The difference in the change in intensity of headache, as measured on an 11-point Numerical Rating Scale (NRS) where 0 means no pain and 10 worst pain imaginable
Onset of headache | at 30 minutes post-intervention and on the morning of day 1, 3, 7, and 14 post-intervention
  The time of onset or worsening of headache when positioned in a sitting position
Sitting endurance | at 30 minutes post-intervention and on the morning of days 1, 3, 7, and 14 post-intervention (in minutes
  The duration of tolerance in an upright position (i.e. how long the patient can stay in an upright position until the headache becomes unbearable and urges the patient to lie down))
SIH associated central nerve system symptoms, such hearing loss, tinnitus, tremor, balance difficulties | at 30 minutes post-intervention and on days 1, 3, 7, and 14 post-intervention
  To assess the impact of SIH-associated symptoms such as tinnitus, tremor, and balance abnormalities
Level of generalized anxiety | at day 14 post-intervention
  Emotional functioning as measured by the Generalized Anxiety Disorder-7 items (GAD-7)
patient satisfaction | at day 14 post-intervention
  patient impression of change, as measured by the Participant Global Impression of Change (PGIC)
analgesic consumption | daily up to day 14
  Analgesic requirement will be measured daily, by intake frequency and dose of analgesics and average daily oral morphine equivalent (OME) in mg
adverse effects | daily up to day 14
Level of Pain Catastrophizing | at Day 14 post-intervention
  Emotional functioning as measured by the Pain Catastrophizing Scale (PCS)
Level of depression | at Day 14 post-intervention
  Emotional functioning as measured by the Patient Health Questionnaire for Depression-9-items (PHQ-9)

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No